CLINICAL TRIAL: NCT06753773
Title: The Short-term Impact of Different Types of Red Light Therapy on Choroid and Retina
Brief Title: Red Light Therapy: Short-term Choroidal and Retinal Changes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSEARS20240715002
Record Dates: First submitted 2024-11-19; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-11

CONDITIONS: Myopia
Keywords: myopia; red light therapy; choroidal; retinal
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard group (Active Comparator): 15 subjects will be recruited in the Standard group, where participants will use the current standard Repeated Low-Level Red-Light device.
  Interventions: Device: Repeated Low-Level Red-Light
- Other types of red light therapy group (Experimental): These 45 subjects will be randomly assigned into three groups: small circle, medium circle, and annular red light groups without disclosure of their specific group to maintain study blinding.
  Interventions: Device: Repeated Low-Level Red-Light

INTERVENTIONS:
Device: Repeated Low-Level Red-Light — All participants will receive a video guide of the Repeated Low-Level Red-Light device. Eligible subjects will receive daily treatment for 14 days, with each treatment lasting for 3 minutes twice a day, with a minimal interval of 4 hours.

SUMMARY:
This research project is a prospective, randomized controlled trial designed to assess the short-term effects of varied red light therapies on the choroidal and retinal structures in adult myopes. The primary objective is to determine which specific retinal regions or cells are primarily affected by short-term repeated low-level red-light (RLRL) therapy, potentially inducing choroidal thickening. The secondary objective is to assess the safety of different types of red light therapy in adult myopes.

The study will enroll 45 myopic adults aged 18-40 years old as participates. They will be randomly assigned into three RLRL groups: small circle (d=0.30mm), medium circle (d=0.50mm), and annular groups (an inner diameter of 0.50 mm and an outer diameter of 0.70mm) without disclosure of their specific group to maintain study blinding. The groups are differentiated by the size and shape of the light spots formed on the retina but with the same power (0.15 mW with a 4 mm pupil size). The Eyerising Myopia Management Device, modified for this study, will be used to administer RLRL with three different spot patterns, adhering to safety standards to minimize risk and ensure participant safety.

Before the treatment, baseline data will be collected from each participant. Baseline assessments will consist of demographics information, visual acuity checks, axial length measurements, subjective refraction, slit-lamp examinations, adaptive optics imaging, optical coherence tomography and angiography (OCT & OCTA), posterior blood flowgraphy, electroretinography (ERG), and the Flicker-plus test. Then participants will undergo daily treatments for 14 days, using the therapy settings of the group to which they have been assigned. The treatment will last for 3 minutes twice a day, with a minimal interval of 4 hours. During the 14-day study period, participants will undergo daily assessments by a series of ophthalmic examinations.

Outcomes measured will track changes in choroidal thickness, electrical activity of the retina, axial length, and best corrected visual acuity, alongside other image reports such as adaptive optics imaging, posterior blood flowgraphy and OCT & OCTA scans.

This study addresses the gaps in understanding how RLRL therapy affects myopia and aims to identify the retina's high-response areas to red light. By doing so, it hopes to minimize unnecessary exposure and potential damage, enhancing the safety and effectiveness of the therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 40 years.
2. Myopic spherical equivalent refraction (SER) between -1.00D to -6.00D in both eyes.
3. Best corrected visual acuity (BCVA): 20/20 or greater.
4. Informed consent for participation.

Exclusion Criteria:

1. Anisometropia greater than 1.50D.
2. Ophthalmic diseases other than refractive errors, including but not limited to strabismus and binocular vision abnormalities in either eye.
3. Systemic diseases (e.g., endocrine, cardiac diseases) and developmental abnormalities.
4. Inability to attend regular follow up assessment.
5. Undergo RLRL therapy in the past 6 months
6. Contraindications to RLRL therapy.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-22 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in choroidal thickness measured by OCT | Choroidal thickness will be measured every day from enrollment to the end of treatment at 2 weeks.
  The change in choroidal thickness (ChT) after 14-day of repeated low-level red-light therapy in adult myopes. OCT and OCTA imaging will be performed using the ultra-wide field swept-source OCT/A system (VG200). The macula was scanned using the 12-line radial scan pattern with a resolution of 1024 × 12. Each image will cover an area of 12 × 9 mm centered on the fovea with an average of 4 consecutive scan overlaps. ChT is defined as the perpendicular distance between the outer choroid-sclera margin and the retinal pigment epithelium-Bruch's complex. The average ChT of the whole ETDRS 9 grid and central ChT (an area centered on the fovea with a diameter of 1 mm) was calculated with the built-in software. The VG200 device has been acquired by our team and is available for use.

SECONDARY OUTCOMES:
Change in electrical activity of the retina measured by ERG | ERG will be carried out on the 7th and 14th days of the study
  A standard full-field ERG and mfREG will be conducted. The full-field ERG includes Dark-adapted 0.01 ERG, Dark-adapted 3.0 ERG, Light-adapted 3.0 ERG, and 30 Hz Flicker ERG. Prior to testing, patients will undergo appropriate dark adaptation for 20 minutes to ensure accurate results for the dark-adapted tests.
Change in axial length (AL) measured by IOL Master | AL will be taken every day from enrollment to the end of treatment at 2 weeks.
  IOL Master will be used to measure the AL of both eyes. Five measurements will be taken for each eye. The AL measurement will be based on the mean of these five values if the desired precision (≤0.05 mm) is achieved.
Change in best corrected visual acuity (BCVA) | BCVA will be taken every day from enrollment to the end of treatment at 2 weeks.
  An Early Treatment Diabetic Retinopathy Study (ETDRS) chart (Precision Vision, Villa Park, Illinois, USA) with standard illumination will be used to measure distance visual acuity. Visual acuity measurement is performed at a distance of 4 meters. BCVA will be measured.
Change in adaptive optics imaging | Adaptive optics imaging assessment will be carried out on the 7th and 14th days of the study.
  The adaptive optics retinal camera rtx1 system (Imagine Eyes) will be employed for high-resolution imaging of cones and rods cells.
Change in optical coherence tomography angiography (OCTA) scan | OCTA assessment will be taken every day from enrollment to the end of treatment at 2 weeks.
  OCT and OCTA imaging will be performed using the ultra-wide field swept-source OCT/A system (VG200). The macula was scanned using the 12-line radial scan pattern with a resolution of 1024 × 12. Each image will cover an area of 12 × 9 mm centered on the fovea with an average of 4 consecutive scan overlaps.
Change in posterior blood flowgraphy | The posterior blood flowgraphy will be taken every day from enrollment to the end of treatment at 2 weeks.
  The Laser Speckle Flowgraphy system (LSFG-NAVI) will be utilized to assess blood flow in the posterior segment of the eye. This method involves capturing and analyzing dynamic changes in speckle patterns created by laser light reflecting off moving blood cells, specifically targeting the retinal and choroidal blood flow. The LSFG-NAVI device has been acquired by our team and is available for use.
Change in flicker-plus test | Flicker-plus test will be carried out on the 7th and 14th days of the study
  The Flicker-plus test, part of the AVOT system, quickly identifies losses in rod and cone photoreceptors without extensive dark adaptation by measuring flicker modulation thresholds (FMTs) at five key central vision points. Adaptation times are minimal-15 seconds for cones and 90 seconds for rods. The test protocol follows the methodologies established by Amithavikram et al.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No